CLINICAL TRIAL: NCT04674527
Title: A Pilot Study of Elemene Injectable Emulsion in Treating Patients With Refractory Glioblastoma
Brief Title: Pilot Study of Elemene in Treating Patients With Refractory Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU-RCT-ELEMENE
Record Dates: First submitted 2020-11-17; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Refractory Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — elemene; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Maintenance chemotherapy with TMZ will be administered at 150-200 mg/m2/day for 5 days in each 28-day cycle.And elemene injectable emulsion will be given for 80 -120 ml/day in each 14-day cycle or 21-day cycle.
  Interventions: Drug: Elemene; Drug: Temozolomide
- contral group (Experimental): Maintenance chemotherapy with TMZ will be administered at 150-200 mg/m2/day for 5 days in each 28-day cycle.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Elemene — Elemene injectable emulsion will be given for 80 mg/day in each 14-day cycle.
  Other Names: elemene injectable emulsion
  Arms: experimental group
Drug: Temozolomide — Maintenance chemotherapy with TMZ will be administered at 150 mg/m2/day for 5 days in each 28-day cycle.
  Other Names: TMZ

SUMMARY:
This is a pilot phase I study to evaluate the safety and efficacy on elemene injectable emulsion in treating patients with glioblastoma. Elemene, isolated from the Chinese medicinal herb Curcuma wenyujin, was shown to exhibit antitumor activity in human and murine tumor cells in vitro and in vivo.Elemene injectable emulsion against malignant tumors was low. Therefore, the effect of Elemene injectable emulsion being used in clinical settings needs to be confirmed by further RCTs.

DETAILED DESCRIPTION:
Background

* Elemene, isolated from the Chinese medicinal herb Curcuma wenyujin, was shown to exhibit antitumor activity in human and murine tumor cells in vitro and in vivo
* The study shows that the methodological quality of RCTs of Elemene injectable emulsion against malignant tumors was low. Therefore, the effect of Elemene injectable emulsion being used in clinical settings needs to be confirmed by further RCTs

Objectives

* To evaluate the safety of Elemene injectable emulsion to treat Refractory Glioblastoma with TMZ
* To evaluate the efficacy of Elemene injectable emulsion to treat Refractory Glioblastoma with TMZ

Design

This clinical trail is a randomized controlled trial.In control group,patients will receive TMZ-chemotherapy.In experimental group,patients will receive elemene injectable emulsion and TMZ-chemotherapy at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; Male or Female.
2. Relapsed/refractory disease confirmed by radiographic evidence after standard therapy.
3. KPS ≥ 60
4. ≥ 8 weeks after completion of front-line radiation therapy
5. ≥ 6 weeks after completion of nitrourea chemotherapy
6. ≥ 14 days after completion of Temozolomide or other chemotherapy
7. 2 weeks of wash-out time after completion of targeted therapy with related adverse events (AE) on baseline
8. White blood cell count (WBC) ≥ 3.0 x 109/L; peripheral blood lymphocyte (PBL) ≥ 25%.
9. Echocardiographic assessment of left ventricular ejection fraction (LVEF) ≥ 40% within 1 month of enrollment.
10. Patients must be able to understand the investigational nature of the study and provide informed consent.

Exclusion Criteria:

1. Those who are allergic constitution, or have contraindications to CT and MRI1 contrast agents.
2. Those who plan to receive any other anti-tumor treatment during the trial.
3. Combined with serious primary diseases of cardiovascular, liver and kidney, and liver function (ALT, AST, Y-GT) exceeding 1.5 times of the upper limit: BUN or Cr exceeding 1.5 times of the upper limit of normal value.
4. Patients with other malignant tumors.
5. Those with active infections, etc.
6. Suspected or confirmed a history of alcohol and drug abuse.
7. Psychiatric illness, intellectual and language disabilities that compromise the informed consent process, at the discretion of the investigator.
8. Women who are pregnant or nursing.
9. Women of childbearing age who refuse to contraception.
10. Active participation in another clinical treatment trials.
11. According to the judgment of the investigator, other conditions that the plan cannot be followed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
overall survival(OS) | 2 years.
  Kaplan Meier methods will be used to estimate median OS.
progression-free survival(PFS) | 2 years.
  Kaplan Meier methods will be used to estimate median PFS. Progression is defined by Response Assessment in Neuro-Oncology (RANO) criteria.

SECONDARY OUTCOMES:
objective response rate(ORR) | 2 years,up to 15 years if necessary.
  Objective Response Rate (ORR) will be assessed by comparison with baseline magnetic resonance imaging by RANO.
complete response(CR) | 2 years,up to 15 years if necessary.
  Complete Response (CR) is disappearance of all measurable and non-measurable disease for at least 4 weeks.
partial response | 2 years,up to 15 years if necessary.
  Partial Response (PR) is ≥ 50% decrease in lesions for at least 4 weeks.
duration of response | 2 years,up to 15 years if necessary.
  Duration of Response (DOR) is the time between the initial response to the treatment and subsequent disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Zhang, MD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No